CLINICAL TRIAL: NCT06708091
Title: A Retrospective Chart Review Combined With a Prospective Cross-sectional Survey and Interviews on Patients With Type 2 Diabetes Mellitus to Assess Effectiveness of Adding SodiumGlucose Co-transporter 2 Inhibitor to Gliclazide Modified Release
Brief Title: Real-world Clinical Effectiveness and Patient Insight Associated With Adding Sodium Glucose Co-transporter 2 Inhibitor to Gliclazide Modified Release
Acronym: ADD2DIA
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-05762-005
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
Keywords: observational; HbA1c; type 2 diabetes; gliclazide MR; SGLT2i; gliclazide MR combined to SGLT2i; retrospective; chart review
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- population description: adult patients with T2DM who initiated add-on SGLT2i treatment to gliclazide MR 60 mg, in routine practice

SUMMARY:
The study objectives are to assess over the gliclazide MR-SGLT2i combined treatment course in patients with T2DM adding SGLT2i to gliclazide MR-based therapy.

The primary objective is to determine the effectiveness of adding SGLT2i to gliclazide MR-based therapy in patients with T2DM, as measured by HbA1c changes.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with T2DM for at least two years prior to index date
* Patient aged ≥18 years at the index date
* Patient naïve to SGLT2i prior to index date
* Patient treated with gliclazide MR at a minimum daily dose of 60 mg at the index date
* Starting treatment with SGLT2i added to gliclazide MR based therapy, during the eligibility period, with a minimum of 60 days of combined gliclazide MR-SGLT2i treatment
* Presence of at least two assessments of HbA1c laboratory test results from the medical records

Exclusion Criteria:

* Diagnosis of diabetes other than T2DM (e.g., type 1, gestational) at index date
* Use of antidiabetic drugs other than those permitted by the inclusion criteria, at index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female who are treated by Gliclazide MR 60 at index date and who started with SGLT2i added to gliclazide MR with a minimum of 60 days of these combined treatments during the eligibility period
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of adding SGLT2i to gliclazide MR | from index date (date of SGLT2i adding to gliclazide MR) to discontinuation of the combination (at least 2 months) or date of data collection initiation during the eligibility period, loss to follow-up, or death, whichever occurs first (approx 2 months)
  To determine the effectiveness of adding SGLT2i to gliclazide MR-based therapy in patients with T2DM, as measured by HbA1c changes (in %)

CONTACTS AND LOCATIONS:
Locations (1):
- Servier Affaires Médicales, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreira RO, Nicodemus NA Jr, Comlekci A, Yu M, Almalki MH. ADD2Dia: Real-World Clinical Effectiveness of Adding a Sodium-Glucose Cotransporter 2 Inhibitor to Gliclazide-Based Therapy in Type 2 Diabetes. Adv Ther. 2025 Dec;42(12):6295-6309. doi: 10.1007/s12325-025-03394-2. Epub 2025 Nov 1. PMID 41175321